CLINICAL TRIAL: NCT05005923
Title: Effect of Non-Surgical Periodontal Therapy on Salivary and Serum Biomarkers in Stage III Grade B and C Periodontitis
Brief Title: Effect of Periodontal Therapy on Biomarkers in Periodontitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAG-A-230119-0014
Record Dates: First submitted 2021-07-29; First posted 2021-08-16 (Actual); Last update posted 2021-08-16 (Actual); Status verified 2021-08

CONDITIONS: Periodontal Health; Periodontitis
Keywords: periodontitis; periodontal treatment
MeSH Terms: conditions — Periodontitis | interventions — Root Planing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Periodontal healthy (No Intervention)
- Periodontitis Stage III Grade B (Active Comparator): The patients were subjected to quadrant-wise full-mouth subgingival scaling and root planning under local anesthesia. The entire non-surgical periodontal treatment of periodontitis groups was completed in a total of 4 sessions in two weeks.
  Interventions: Procedure: Non-surgically performed scaling and root planing
- Periodontitis Stage III Grade C (Active Comparator): The patients were subjected to quadrant-wise full-mouth subgingival scaling and root planning under local anesthesia. The entire non-surgical periodontal treatment of periodontitis groups was completed in a total of 4 sessions in two weeks.
  Interventions: Procedure: Non-surgically performed scaling and root planing

INTERVENTIONS:
Procedure: Non-surgically performed scaling and root planing — Treatment of patients with periodontitis was performed using manual and ultrasonic instruments.
  Arms: Periodontitis Stage III Grade B; Periodontitis Stage III Grade C

SUMMARY:
The present study aimed to assess the effect of non-surgical periodontal treatment on serum and salivary MMP-8, MAF, MIP-1α, M-CSF, and IL34 levels in periodontitis stage III grade B (P-III-B) and C (P-III-C) patients. 20 periodontally healthy, 20 P-III-B and 25 P-III-C participants were enrolled. At baseline, serum and saliva samples were collected and the whole mouth clinical periodontal parameters were recorded. Periodontitis patients received non-surgical periodontal treatment. Clinical parameters were re-measured and samples were re-collected at 1 and 3 months after treatment. Serum and salivary MMP-8, MAF, MIP-1α, M-CSF, and IL34 levels were analyzed by ELISA. Data were analyzed using appropriate statistical tests.

DETAILED DESCRIPTION:
Periodontal disease is an inflammatory process that can result in tooth loss and also is considered a modifying factor for systemic health. Matrix metalloproteinase (MMP)-8 is the major collagenase of periodontal tissue breakdown. Macrophage-activating factor (MAF) can activate macrophages. M-CSF is known to modulate disease and inflammation and to play an important role in bone destruction. IL-34 shares vital functions of M-CSF, and manages myeloid cell survival, differentiation, and proliferation.

This study is the first controlled clinical study that examines the levels of MIP-1α, MAF, MMP-8, M-CSF, IL-34 in saliva and serum in two different periodontitis, and evaluates the situation before and after the treatment. The first hypothesis of this study; in periodontitis group, salivary and serum MIP-1α, MAF, MMP-8, M-CSF, IL-34 levels will be high, in contrast to the periodontal healthy group. The second hypothesis of this study is that after periodontal treatment, saliva and serum MIP-1α, MAF, MMP-8, M-CSF, IL-34 levels will decrease. Based on these hypotheses, the aim of the study is; to compare the levels of MIP-1a, MAF, MMP-8, M-CSF, IL-34 in saliva and serum of healthy controls, P-III-B, and P-III-C subjects and to evaluate the effect of periodontal treatment.

A total of 65 systemically healthy patients; 20 periodontally healthy, 20 P-III-B, 25 P-III-C were included in this study. The whole mouth clinical periodontal examination included measurement of probing depth (PPD), clinical attachment level (CAL), presence of bleeding on probing (BOP), gingival index (GI), and plaque index (PI) at 6 sites per tooth, except the third molars. The presence and type of the alveolar bone loss were assessed on the digital panoramic radiograph in each participant, which was supplemented with periapical radiographs if necessary.

Periodontal status of each patient was evaluated by a single calibrated periodontists with a manual probe. The diagnosis of periodontitis or periodontally health was determined according to the 2017 World Workshop on Classification of Periodontal and Peri-Implant Diseases and Conditions. Periodontally healthy individuals (n=20) in the control group had no sites with PD >3 mm and CAL >2 mm and also no radiographic evidence of alveolar bone loss. BOP was <10% in the whole mouth. Healthy group also exhibited no history of periodontitis. The periodontitis stage III patients had a minimum three teeth apart from the first molars and incisors showing CAL ≥5 mm and PD ≥6 mm and showed no>4 teeth loss because of periodontitis. Radiographic bone loss extending from coronal to middle third or beyond. Radiographic bone loss was determined from the tooth showing the most severe bone loss as a percentage of root length. If the values of bone loss %/age were between 0.25 and 1.0, the patients were assigned to grade B (n=20). If higher than 1.0, the patients were assigned to grade C (n=25)

Treatment

The recruited periodontitis patients received conventional quadrant scaling and root planning (SRP) under local anesthesia in a total of 4 sessions in two weeks. SRP was performed by the same periodontist using ultrasonic inserts and manual periodontal curettes. Re-evaluations were performed at 1 and 3 months following the completion of the SRP. No periodontal intervention was carried out in the periodontally healthy controls.

Saliva and Serum Sampling A total of 5 mL of unstimulated whole saliva was collected by passive drool method between 9:00 and 10:00 am. The participants were advised to avoid food consumption for three hours before sample collection. The participants were seated upright and saliva was collected over a period of 5 minutes with instructions to pool saliva in the floor of the mouth and passively drool it into a sterile glass beaker. Then saliva samples are immediately transferred to a 2 mL polypropylene tube and stored at -80°C. A total of 5 mL of blood was collected from the antecubital fossa by venepuncture method. Serum was isolated from the blood by centrifuging at 5000 rpm for 10 minutes followed by its rapid transfer to a sterile polypropylene tube and storage at -80°C.

Biomarker Immunoassays Saliva and serum samples were thawed on ice. The saliva samples were centrifuged at 5.000 rpm for 15 minutes at room temperature, and supernatants were immediately used for assays. Serum and salivary samples of MMP-8 , M-CSF*, MIP-1α*, MAF , IL-34 in were measured by ELISA using commercial kits.

Statistical Analysis All statistical analyses were carried out with the standard statistical software package. For the intra-group comparisons, if the data were not normally disturbed, Friedman test and the Dunn test with the Bonferroni correction were used to analyze the change between baseline and 1 month and 3 months after treatment. For inter-group comparisons, Mann-Whitney U test for normally and non-normally disturbed data. The Spearman's rank correlation test was used to detect the correlations of biochemical parameters with clinical parameters and each others in diseased group before and after treatment. All tests were performed at significance level of P <0.05.

ELIGIBILITY:
Inclusion Criteria:

1. systemically healthy and non-smoker individuals
2. having ≥20 teeth present (except third molars)
3. individuals with periodontally healthy, periodontitis stage III grade B and C diagnoses

Exclusion Criteria:

1. having any diagnosed medical disorders such as diabetes mellitus, cardiovascular diseases, rheumatoid arthritis, immunological and mucocutaneous diseases
2. usage of antibiotics, non-steroidal anti-inflammatory drugs and immunosuppressive agents within the past 6 months
3. having any non-inflammatory destructive periodontal disease
4. nonsurgical/surgical periodontal therapy received in the past year
5. pregnant/ lactating/ postmenopausal females.

Ages: 23 Years to 51 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2019-01-23 (Actual); Primary Completion 2020-07-24 (Actual); Study Completion 2020-07-24 (Actual)

PRIMARY OUTCOMES:
Salivary MMP-8 (ng/ml) level | baseline to 1 month and 3 months after treatment
  change in salivary MMP-8 levels from baseline to 1 month and 3 months after treatment
Salivary MAF (ng/ml) level | baseline to 1 month and 3 months after treatment
  change in salivary MAF levels from baseline to 1 month and 3 months after treatment
Salivary MIP-1α (pg/ml) level | baseline to 1 month and 3 months after treatment
  change in salivary MIP-1α levels from baseline to 1 month and 3 months after treatment
Salivary M-CSF (pg/ml) level | baseline to 1 month and 3 months after treatment
  change in salivary M-CSF levels from baseline to 1 month and 3 months after treatment
Salivary IL-34 (pg/ml) level | baseline to 1 month and 3 months after treatment
  change in salivary M-CSF levels from baseline to 1 month and 3 months after treatment

SECONDARY OUTCOMES:
Serum MMP-8 (ng/ml) level | baseline to 1 month and 3 months after treatment
  change in serum MMP-8 levels from baseline to 1 month and 3 months after treatment
Serum MAF /ng/ml) level | baseline to 1 month and 3 months after treatment
  change in serum MAF levels from baseline to 1 month and 3 months after treatment
Serum MIP-1α (pg/ml) level | baseline to 1 month and 3 months after treatment
  change in serum MIP-1α levels from baseline to 1 month and 3 months after treatment
Serum M-CSF (pg/ml) level | baseline to 1 month and 3 months after treatment
  change in serum M-CSF levels from baseline to 1 month and 3 months after treatment
Serum IL-34 (pg/ml) level | baseline to 1 month and 3 months after treatment
  change in serum IL-34 levels from baseline to 1 month and 3 months after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University, Faculty of Dentistry, Department of Periodontology, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided